CLINICAL TRIAL: NCT00330265
Title: A Prospective, Randomized, Controlled, Unmasked, Multiple Treatment, Multi-Center Clinical Trial to Evaluate the Efficacy and Safety of an Interactive Wound Dressing Containing Cultured Keratinocytes Versus Conventional Wound Therapy for the Treatment of Diabetic Foot Ulcers
Brief Title: Safety and Efficacy Study of an Interactive Wound Dressing (KC002) for the Treatment of Diabetic Foot Ulcers
Acronym: KC-002PT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: KeraCure (Industry)
Responsible Party: KeraCure, KeraCure
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCT 20051320
Record Dates: First submitted 2006-05-24; First posted 2006-05-26 (Estimated); Last update posted 2008-08-26 (Estimated); Status verified 2008-08

CONDITIONS: Foot Ulcer; Diabetes
MeSH Terms: conditions — Foot Ulcer; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): KC-002
  Interventions: Device: KC-002
- 2 (Other): Conventional Wound Therapy
  Interventions: Other: Conventional Wound Therapy

INTERVENTIONS:
Device: KC-002 — Determine the safety and effectiveness of a device (the KC-002 interactive wound dressing) in the promotion of healing in diabetic foot ulcers as compared with a conventional wound therapy regimen for subjects with Type 1 or Type 2 diabetes mellitus.
  Arms: 1
Other: Conventional Wound Therapy — Normal Saline Dressings
  Arms: 2

SUMMARY:
The objective of this study is to determine the safety and effectiveness of a device (the KC-002 interactive wound dressing) in the promotion of healing in diabetic foot ulcers as compared with a conventional wound therapy regimen for subjects with Type 1 or Type 2 diabetes mellitus.

This is a prospective, randomized, multi-center, unmasked, controlled study. All patients will receive care for the diabetic foot ulcer during the study.

Participation in the study is for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

Participants included in the study must:

* Have Type 1 or Type 2 diabetes mellitus
* Have a diabetic foot ulcer on the bottom of the foot or heal which has been present for three (3) weeks but less than two (2) years and is sufficient size to qualify for the study
* Be able to visit the study doctor regularly for 24 weeks

Exclusion Criteria:

Participants may not be included if:

* The diabetic foot ulcer is infected
* They have poor circulation in their study foot
* Cannot or will not wear a special boot to take pressure off the study ulcer
* They have certain other diseases or laboratory values which are not within a specified range

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-01; Primary Completion 2009-03 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Percent of subjects achieving complete or (100%) study wound closure by week 12 after initial treatment | 12 weeks

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Institute for Advanced Wound Care at Baptist Medical Center South, Montgomery, Alabama
  - HOPE Research Institute, Phoenix, Arizona
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Roy Kroeker, DPM, Fresno, California
  - Felix Sigal, DPM, Los Angeles, California
  - Bay Area Foot Care, San Francisco, California
  - North American Center for Limb Preservation, New Haven, Connecticut
  - Georgetown University / Wound Healing Center, Washington D.C., District of Columbia
  - Doctor's Research Network, South Miami, Florida
  - Medical Associates, Clinton, Iowa
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Preston Family Building, Boston, Massachusetts
  - Foot Healthcare Associates, PC, Livonia, Michigan
  - St. Vincent Health Center Wound Clinic, Erie, Pennsylvania
  - Pivotal Clinical Research, Souderton, Pennsylvania
  - Warren General Hospital Wound Clinic, Warren, Pennsylvania
  - Martin Foot and Ankle, York, Pennsylvania
  - San Antonio Podiatry Associates, PC, San Antonio, Texas
  - Pharmaceutical Research Organization, Bountiful, Utah
  - Dixie Regional Medical Center's Wound Clinic, St. George, Utah
  - Central Washington Podiatry Service, Yakima, Washington